CLINICAL TRIAL: NCT04520607
Title: A Long-Term Extension Study Evaluating the Safety and Efficacy of Lorecivivint in Subjects With Osteoarthritis of the Knee
Brief Title: A Long-Term Safety and Efficacy Study of Lorecivivint in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SM04690-OA-07
Record Dates: First submitted 2020-08-14; First posted 2020-08-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
Keywords: SM04690; Wnt pathway inhibitor; osteoarthritis; Biosplice Therapeutics, Inc.; Samumed; lorecivivint
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — lorecivivint

STUDY DESIGN:
Who Masked: Participant
Masking Description: Note: The first 48 weeks will be single-blind and placebo-controlled while the remainder of the study will be open-label and uncontrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Subjects assigned to this arm will receive one intra-articular injection of 0.07 mg lorecivivint in 2 ml vehicle (same treatment as in the parent-study) into their target knee (the same target knee injected in the parent study); performed on Day 1, at Week 48 and every 52 weeks thereafter.
  Interventions: Drug: Lorecivivint
- Arm 2 (Experimental): Subjects assigned to this arm will receive one intra-articular injection of 0 mg lorecivivint in 2 ml vehicle (same treatment as in the parent-study) into their target knee (the same target knee injected in the parent study) on Day 1, followed by one intra-articular injection of 0.07 mg lorecivivint in 2 ml vehicle at Week 48 and every 52 weeks thereafter.
  Interventions: Drug: Placebo; Drug: Lorecivivint

INTERVENTIONS:
Drug: Placebo — Healthcare professional-administered intra-articular injection of vehicle.
  Other Names: Vehicle
  Arms: Arm 2
Drug: Lorecivivint — Healthcare professional-administered intra-articular injections of lorecivivint.
  Other Names: SM04690

SUMMARY:
This study is designed as a long-term extension to the Phase 3 parent-study SM04690-OA-11. It aims to evaluate the safety and efficacy of long-term use of lorecivivint (LOR) in subjects with knee osteoarthritis (OA). The first 48 weeks will be single-blind and placebo-controlled while the remainder of the study will be open-label and uncontrolled. Subjects must enroll no later than 6 weeks following completion of the parent-study.

DETAILED DESCRIPTION:
At the first visit (Day 1), all subjects will complete Patient Acceptable Symptom State (PASS) and pain Numeric Rating Scale (NRS) assessments and then receive a blinded study injection into their target knee (the same target knee injected in the parent study), with subjects receiving the same treatment (either 0.07 mg LOR or placebo) as they received in the parent study. Subjects will have clinic visits for pain and function assessments, collection of adverse events, and knee radiographs. At Week 48, all subjects, regardless of previous treatment, will receive an injection of 0.07 mg LOR into their target knee. Subjects will receive injections of 0.07 mg LOR into their target knee every 52 weeks thereafter until end of study.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of the Samumed study SM04690-OA-11
2. Compliance with procedures in study SM04690-OA-11, in the opinion of the Investigator
3. Fully understanding study requirements and willingness to comply with study visits and assessments
4. Understanding and signing of the informed consent form (ICF) prior to any study-related procedures

Exclusion Criteria:

1. Any condition that, in the opinion of the Investigator, constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct, or evaluation
2. Any contraindications for an intra-articular (IA) injection in the target knee in the opinion of the Investigator
3. Any known reason identified by the Investigator or Sponsor that the subject may not be compliant with study visits or may no longer be an appropriate candidate for the study (e.g. planned major surgery, knee replacement during the parent study, planning to move away from the research site, or initiation of a prohibited concomitant medication including, but not limited to, IA injection of glucocorticoids, hyaluronic acid derivatives, platelet-rich plasma, stem cell therapies, or other agents with therapeutic intent into the target knee)
4. Participation in a clinical research trial (other than the prior SM04690-OA-11 study) that included the receipt of an investigational product (IP) or any experimental therapeutic procedure within 12 weeks before any study injection, or planned participation in any such trial
5. Current or pending disability claim, workers' compensation, or litigation(s) that may compromise response to treatment
6. Pregnant women, breastfeeding women, and women who are not post-menopausal (defined as 12 months with no menses without an alternative medical cause) or permanently surgically sterile (includes hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) who have a positive or indeterminate pregnancy test result at Visit 1E (Day 1)
7. Women who are not post-menopausal or permanently surgically sterile who are sexually active, and who are not willing to use birth control (as outlined in the protocol) during the study period

Ages: 41 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Primary Safety Outcome: Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Visit 1E (Day 1) through Visit 3E (Week 48)
  AEs that occur during the study will be recorded, and ongoing AEs at the end of the parent-study will continue to be monitored. All AEs will be evaluated for severity, seriousness and causal relationship to study medication.
Primary Efficacy Outcome: Change from parent-study baseline medial joint space width (mJSW) in the target knee | Parent-study baseline; Visit 3E (Week 48)
  Change from parent-study baseline in mJSW as documented by radiograph (X-ray) of the target knee

SECONDARY OUTCOMES:
Change from parent-study baseline OA pain in the target knee | Parent-study baseline; Visit 2E (Week 24)
  Change from parent-study baseline OA pain in the target knee as assessed by the weekly averages of daily pain Numeric Rating Scale (NRS). The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.
Change from parent-study baseline OA function in the target knee | Parent-study baseline; Visit 2E (Week 24)
  Change from parent-study baseline OA function in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numeric Rating Scale (NRS 3.1) physical functioning subscore (WOMAC Function). The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore ranges from 0 to 170.
Change from parent-study baseline OA pain in the target knee | Parent-study baseline; Visit 3E (Week 48)
  Change from parent-study baseline OA pain in the target knee as assessed by the weekly averages of daily pain Numeric Rating Scale (NRS). The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 represents the worst possible pain.
Change from parent-study baseline OA function in the target knee | Parent-study baseline; Visit 3E (Week 48)
  Change from parent-study baseline OA function in the target knee as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numeric Rating Scale (NRS 3.1) physical functioning subscore (WOMAC Function). The WOMAC is a widely-used, proprietary outcome measurement tool used by health professionals to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions), and physical functioning (17 questions) of the joints. Each question is measured on a scale from 0 (lowest pain/lowest stiffness/highest function) to 10 (highest pain/highest stiffness/lowest function). The WOMAC Function subscore ranges from 0 to 170.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Simsek, MD, Study Director — Biosplice Therapeutics, Inc.
Locations (42):
- United States (42):
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Pomona, California
  - Research Site, San Diego, California
  - Research Site, Thousand Oaks, California
  - Research Site, Denver, Colorado
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Port Orange, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Newnan, Georgia
  - Research Site, Woodstock, Georgia
  - Research Site, Gurnee, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Valparaiso, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Bay City, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Hazelwood, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Omaha, Nebraska
  - Research Site, Hartsdale, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Fort Mill, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Carrollton, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Draper, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No